CLINICAL TRIAL: NCT05334576
Title: Study of Crizanlizumab for Prevention of Silent Cerebral Infarcts in SCA Novartis Investigator Initiated Trial: CSEG101AUS12T
Brief Title: Study of Crizanlizumab for Prevention of Silent Cerebral Infarcts in SCA
Acronym: CRIZ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Andria Ford (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Andria Ford, Principal Investigator, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CSEG101AUS12T
Record Dates: First submitted 2021-11-30; First posted 2022-04-19 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — crizanlizumab

STUDY DESIGN:
Intervention Model Description: Crizanlizumab (SEG101) at 5.0 mg/kg dose administered over two years per standard of care in patients with sickle cell disease and silent cerebral infarcts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm: Crizanlizumab (Other): Single-arm: Patients with sickle cell disease and increased risk of silent cerebral infarcts
  Interventions: Other: Crizanlizumab

INTERVENTIONS:
Other: Crizanlizumab — Crizanlizumab 5.0 mg/kg infusions will be administered over 24 months

SUMMARY:
In this prospective, single-arm, open-label, imaging and treatment study, the investigator will test the hypothesis that crizanlizumab will prevent the progression of silent cerebral infarcts in patients with sickle cell disease. Study participants will undergo brain MRI before initiation of crizanlizumab and at 6 and 30 months after starting crizanlizumab infusions. The crizanlizumab cohort will be compared to a matched, observational cohort of patients not receiving crizanlizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants age 16 and older
2. Sickle cell disease with confirmation of HbSS, HbSBthal0, HbSC, or HbS thal+ genotype
3. Per patient's sickle cell provider, patient has an increased risk of a silent cerebral infarcts according to one of the following criteria:

   1. Silent cerebral infarcts visualized on FLAIR MRI within previous two years
   2. Intracranial or extracranial cervical artery vasculopathy
   3. History of overt ischemic or hemorrhagic stroke and Intolerance and/or failure of other therapies to prevent cerebral infarction
   4. Increased severity of sickle cell disease including having between 2 and 10 sickle cell-related pain crises within the preceding 12 months as determined by medical history or by patient's recall (crises should include the occurrence of appropriate symptoms, a visit to a specific medical facility and/or health care professional, and receipt of pain medication).
   5. Increased risk deemed by other objective laboratory and/or imaging results which have been associated with increased risk of cerebral infarction
4. Provide written informed consent.
5. Normal hematologic function defined as: WBC > 4x10^9 / L, ANC >1.5x10^9 / L and platelets > 100x10^9 / L
6. Females of childbearing potential (FCBP) must agree to refrain from becoming pregnant while on crizanlizumb and for 3 months after discontinuation from crizanlizumab, and must agree to use adequate contraception including hormonal contraception, (i.e. birth control pills, etc.), barrier method contraception (i.e. condoms), or abstinence during the time-frame

Exclusion Criteria:

1. Current chronic transfusion therapy
2. Planning for hematopoietic stem cell transplant or cerebral revascularization procedure
3. Use of other investigational drug within one year of study participation
4. Other medical/neurological/social/substance abuse history that would alter brain MRI findings prospectively
5. Inability to return for follow-up
6. Contraindication to MRI
7. Acute bacterial, fungal, or viral infection
8. Known HIV, untreated latent tuberculosis (TB), or active hepatitis B or C infection or zoster
9. Pregnant and/or breastfeeding. Negative pregnancy test required prior to starting study treatment.
10. Known hypersensitivity to one or more of the study agents
11. Currently receiving or has received any investigational drugs within the 14 days prior to the first dose of study drug
12. Liver function tests (LFT) higher than 3x the upper limit of normal
13. Treatment with other monoclonal antibody medications within last 30 days
14. Treatment with various forms of anticoagulation within last 30 days, including but not limited to coumadin or direct thrombin inhibitors

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
New or enlarged silent cerebral infarcts | 30 months
  Occurrence of 'new or enlarged' silent cerebral infarcts between the baseline and 30 month follow-up scan.

SECONDARY OUTCOMES:
Infarct Progression | 30 months
  Change in volume of silent cerebral infarcts between the baseline and 30 month follow-up scan.

CONTACTS AND LOCATIONS:
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No